CLINICAL TRIAL: NCT03858257
Title: High Flow Nasal Oxygen During Conscious Sedation in the Cardiac Catheterisation Laboratory: A Randomized Controlled Trial
Brief Title: High Flow Nasal Oxygen During Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Aaron Conway, RBC Chair in Cardiovascular Nursing Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-6343
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia; Cardiac Disease
Keywords: Oxygen; Ventilation; High-flow nasal oxygen; Hypercapnia; Respiratory depression; Respiratory compromise; Carbon dioxide; Transcutaneous carbon dioxide
MeSH Terms: conditions — Heart Diseases; Respiratory Aspiration; Hypercapnia; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal oxygen (Experimental): The gas temperature will commence at the 'High' setting (ranges 30-32º Celsius) and titrated downwards if the patient complains of irritation. The gas flow rate will commence at 30 liters per minute prior to sedation administration and be titrated up to 70 liters per minute as tolerated by the patient after sedation has been administered. The fraction of oxygen in the gas will be commenced at 50% (same as that delivered from 6 liters per minute via facemask) and can be titrated upward according to patient requirements (i.e. increased if there is evidence of hypoventilation, airway obstruction or inadequate oxygenation, decreased during use of diathermy). Anesthesia Assistants at the site will be provided with training in the use of this mode of oxygen delivery prior to study commencement.
  Interventions: Device: High flow nasal oxygen
- Standard oxygenation (Other): Supplemental oxygen through a facemask with the flow rate chosen by the clinician responsible for sedation as per their standard practice. The oxygen flow rate is typically commenced at 6 liters per minute and can be titrated up to 15 liters per minute.
  Interventions: Device: Standard oxygenation

INTERVENTIONS:
Device: High flow nasal oxygen — The Optiflow device (Fisher and Paykel Healthcare, Auckland, New Zealand) will be used.
  Arms: High flow nasal oxygen
Device: Standard oxygenation — Supplemental oxygen through a facemask.
  Arms: Standard oxygenation

SUMMARY:
The primary objective of this study is to test the hypothesis that using high flow nasal oxygen improves ventilation during cardiac implantable electronic device procedures performed with conscious sedation. A randomized controlled trial design will be used with participants randomized in a 1:1 ratio to oxygen supplementation through a standard facemask or high flow nasal oxygen.

DETAILED DESCRIPTION:
High flow nasal oxygen (HFNO) is increasingly regarded as a promising technology for oxygen delivery in critical care and anesthetic management. Although promising, further high-quality studies examining the effects of using HFNO during procedural sedation are required to inform decision-making regarding implementation of this new technology into practice. The 2018 guidelines from the American Society of Anesthesiology stated that there is insufficient evidence regarding which methods of supplemental oxygen administration (e.g., nasal cannula, face mask, or specialized devices such as HFNO) are more effective. This trial will address this limitation in the evidence base specifically in regard to the efficacy of using HFNO during conscious sedation in the cardiac catheterisation laboratory.

ELIGIBILITY:
Inclusion criteria:

1. Adults undergoing an elective cardiac implantable electronic device procedure in the Peter Munk Cardiac Centre Cardiac Cath Labs with conscious sedation administered by an Anesthetic Assistant (de novo and replacement/revision procedures).

Exclusion criteria:

1. Under 16 years of age.
2. Underlying condition requiring chronic oxygen supplementation.
3. Diagnosed respiratory condition with confirmed current hypercapnia.
4. Pre-existing untreated pneumothorax.
5. Transesophageal echocardiography planned for the procedure.
6. Active nasal bleeding.
7. Complete nasal obstruction.
8. Recent upper airway surgery or base of skull fracture.
9. Previous participation in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Peak transcutaneous carbon dioxide (TcCO2) concentration. | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  Continuous measurements will be recorded using the Sentec Digital Monitoring with VSign 2 sensor.

SECONDARY OUTCOMES:
Mean transcutaneous carbon dioxide concentration | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  Continuous measurements will be recorded using the Sentec Digital Monitoring with VSign 2 sensor.
Area under SpO2 90% oxygen desaturation curve | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  Percentage of hemoglobin saturated with oxygen (SpO2) will be measured continuously throughout procedures as part of routine clinical practice through the anaesthetic machine. This is a composite measure comprising the incidence, depth, and duration of oxygen desaturation events. Area under SpO2 90% oxygen desaturation curve is calculated as the difference between the threshold (90%) and actual oxygen saturation (SpO2) summed every second during which oxygen saturation was below threshold.
Adverse sedation events | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  The Anaesthesia Assistant will be asked to complete the Tracking and reporting outcomes of procedural sedation (TROOPS) tool at the end of procedures. Completion of the tool requires identification and description of the adverse event, the intervention, the outcome and the overall severity of the adverse event.
Patient satisfaction with sedation: Iowa Satisfaction with Anesthesia Scale | After the participant has reached phase 2 post-anesthetic recovery. Estimated to be 30 minutes after procedure has finished.
  Iowa Satisfaction with Anesthesia Scale. Score ranges from -3 (worse satisfaction) to +3 (better satisfaction).
Costs associated with oxygen delivery | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  Anesthesia Assistants will document devices used for supplemental oxygen delivery and airway management in both groups as per their usual practice in the anesthesia monitoring system.
Anesthesia Assistant rating of difficulty maintaining the patient's oxygenation status | To be completed as soon as possible after the end of the procedure (within about 5 minutes).
  The Anaesthesia Assistant will be asked to rate their perceived level of difficulty in maintaining oxygenation using a 6-level rating scale with ratings of "extremely difficult", "very difficult", "difficult", "easy", "very easy", "extremely easy".
Anesthesia Assistant rating of difficulty using oxygen delivery device | To be completed as soon as possible after the end of the procedure (within about 5 minutes).
  The Anaesthesia Assistant will be asked to rate their perceived level of difficulty using the oxygen delivery device using a 6-level rating scale with ratings of "extremely difficult", "very difficult", "difficult", "easy", "very easy", "extremely easy".
Patient comfort of oxygen delivery | After the participant has reached phase 2 post-anesthetic recovery. Estimated to be 30 minutes after procedure has finished.
  Participants will be asked to rate at the end of procedures their perceived overall comfort with the oxygen delivery device used during the procedure using a 6-level rating scale with ratings of 'maximal discomfort', 'very uncomfortable', 'uncomfortable', 'comfortable', 'very comfortable' and 'maximal comfort'.
Trajectory of transcutaneous carbon dioxide as a function of time | From the time between first sedative medication administration to the end of the procedure. Estimated duration of procedures is 30 minutes to 120 minutes.
  Continuous measurements will be recorded using the Sentec Digital Monitoring with VSign 2 sensor

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Conway, RN, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study data, participant-level data sets (without identifying information) and code for statistical analyses will be shared in a publicly accessible repository at the time of publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: With publication of results.
Access Criteria: Available through a public repository

REFERENCES:
- [Derived] Conway A, Collins P, Chang K, Kamboj N, Filici AL, Lam P, Parotto M. High flow nasal oxygen during procedural sedation for cardiac implantable electronic device procedures: A randomised controlled trial. Eur J Anaesthesiol. 2021 Aug 1;38(8):839-849. doi: 10.1097/EJA.0000000000001458. PMID 33492872

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT03858257/Prot_SAP_000.pdf